CLINICAL TRIAL: NCT02622932
Title: A Phase 1, Open-label Study to Investigate the Absorption, Metabolism and Excretion of [14C] Anlotinib in Patients With Advanced Cancer Patients
Brief Title: Study to Investigate the Absorption, Metabolism and Excretion of [14C] Anlotinib in Patients With Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-I-R
Record Dates: First submitted 2015-12-02; First posted 2015-12-07 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anlotinib and 14C-labeled Anlotinib (Experimental): each participant will be given a single dose of 14C-labeled gilteritinib.
  Interventions: Drug: Anlotinib and 14C-labeled Anlotinib

INTERVENTIONS:
Drug: Anlotinib and 14C-labeled Anlotinib — oral

SUMMARY:
The purpose of this study is to Investigate the Absorption, Metabolism and Excretion of [14C] Anlotinib in Patients With Advanced Cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* histologically or cytologically confirmed diagnosis of advanced solid tumor (including RCC、NSCLC、STS and CRC)
* failed to the treatment of line 1 or 2
* ECOG PS:0-1,Life expectancy of more than 3 months
* main organs function is normal

Exclusion Criteria:

* prior treatment with Anlotinib or Allergic to drug or its formulation ingredients
* subjects with the gastrointestinal tract, liver and kidney disease of affect drug absorption and metabolism
* CTCAE(4.0) Grade 1 or higher non-remission toxicity induced by any other previous treatments
* patients with pleural effusion or ascites, causing respiratory syndrome (CTCAE Grade 2 or higher dyspnea [Grade 2 dyspnea refers to Shortness of breath with a small amount of activities, affecting Instrumental activities of daily life])
* patients underwent major surgical treatment，open biopsy or significant traumatic injury within 28 days prior to assignment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of 14C-labeled Anlotinib (radioactivity in urine) | up to 10 Days(endpoint when the two consecutive time points of cumulative excretion <1%)
Cumulative excretion of 14C-labeled Anlotinib (radioactivity in feces) | up to 10 Days(endpoint when the two consecutive time points of cumulative excretion <1%)
Excretion rate of 14C-labeled Anlotinib (radioactivity in urine) | up to 10 Days(endpoint when the two consecutive time points of cumulative excretion <1%)
Excretion rate of 14C-labeled Anlotinib (radioactivity in feces) | up to 10 Days (endpoint when the two consecutive time points of cumulative excretion <1%)
Pharmacokinetics of 14C-labeled Anlotinib (Radioactivity in whole blood):Peak Plasma Concentration(Cmax) | up to 10 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak Plasma Concentration(Cmax),Cmax in ng/mL,
Pharmacokinetics of 14C-labeled Anlotinib (Radioactivity in whole blood):Peak time（Tmax） | up to 10 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak time（Tmax）,Tmax in h.
Pharmacokinetics of 14C-labeled Anlotinib (Radioactivity in whole blood):Half life（t1/2） | up to 10 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Half life（t1/2）,t1/2 in h.
Pharmacokinetics of 14C-labeled Anlotinib (Radioactivity in whole blood): Area under the plasma concentration versus time curve (AUC) | up to 10 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Area under the plasma concentration versus time curve (AUC), AUC in ng.h/mL.
Pharmacokinetics of 14C-labeled Anlotinib (Radioactivity in whole blood): Clearance（CL） | up to 10 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Clearance（CL）,CL in L/h.

SECONDARY OUTCOMES:
Metabolite identification of Anlotinib in plasma, urine and feces | up to 10 Days(endpoint when the two consecutive time points of cumulative excretion <1%)

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Bao, Doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided